CLINICAL TRIAL: NCT01405833
Title: Phase 1: A Multi-Centered, Randomized, Blinded, Placebo-Controlled, Serial-Cohort, Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of BG00010 (Neublastin) in Subjects With Sciatica
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Safety of BG00010 (Neublastin) in Subjects With Sciatica.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103NS102
Record Dates: First submitted 2011-07-21; First posted 2011-07-29 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BG00010 (Neublastin) (Experimental): Participants may be randomized to escalating doses of BG00010
  Interventions: Drug: BG00010 (Neublastin)
- Placebo (Placebo Comparator): Participants may be randomised to a matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BG00010 (Neublastin) — Multiple doses, weight-based IV administration
  Arms: BG00010 (Neublastin)
Drug: Placebo — Single dose IV matched placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, and pharmacokinetic (PK) profile of 3 intravenous (IV) injections of BG00010 given on 2 fixed schedules; weekly and as frequently as every 48 hours (but no more than 3 times per week).

Secondary objectives of this study in this study population are to explore the repeated-dose immunogenicity of BG00010 and to explore the potential of BG00010 to reduce pain following multiple-dose administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of unilateral sciatica, determined by the Investigator and as outlined in the protocol. Sciatica symptoms must be present for 3 or more months prior to the Screening Visit.
* Must rate their pain at >/=40 mm on the 100 mm Visual Analog Scale (VAS) of the Short-Form McGill Pain Questionnaire (SF-MPQ)at the Screening and Baseline Visits.

Key Exclusion Criteria:

* History of malignancy or clinically relevant allergies and/or cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (not related to sciatica), dermatologic, rheumatic/joint, psychiatric, renal, and/or other major disease.
* History of severe pain as judged by the Investigator, other than that caused by sciatica during the 3 months prior to Screening Visit.
* Signs or symptoms of peripheral neuropathy, other than symptoms of sciatica during the 3 months prior to Screening Visit.
* Current generalized myalgia
* Serum creatinine >1.5 x upper limit of normal (ULN).
* History of or positive screening test for hepatitis C infection, hepatitis B infection and/or positive for hepatitis B core antibody or positive for human immunodeficiency virus (HIV) antibody. Subjects who are HBsAg negative and HBcAb positive are allowed to participate if they are positive for HBsAb IgG (see the Centers for Disease Control and Prevention's interpretation of the hepatitis B serology panel).
* Treatment with any prescription medication and/or over the-counter products such as herbal supplements, unless the dose has been stable for 2 weeks prior to the Baseline Visit.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants experiencing Adverse Events | Throughout the study period- an expected 15 weeks
Serum drug concentrations of BG00010 as a measure of pharmacokinetics | Throughout the study period- an expected 15 weeks

SECONDARY OUTCOMES:
Presence of anti-BG00010 antibodies in serum | Throughout the study period- an expected 15 weeks
  Assessment of study-treatment-specific safety of BG00010
Change in pain as measured by Likert numerical pain rating scale | Every day for 3 consecutive days prior to baseline throughout the study period
Change in Visual analog Scale (VAS) of the Short-Form McGill Pain Questionnaire (SF-MPQ) | Throughout the study period at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leiden, Netherlands